CLINICAL TRIAL: NCT03756935
Title: Non-invasive and Continuous Detection of Arterial Hypotension Using Photoplethysmographic Signal During Induction of Anaesthesia: Proof of Concept
Brief Title: Early Detection of Intra Operative Hypotension (IOH) During the Induction of General Anaesthesia
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); M3DISIM (Other)
Responsible Party: Principal Investigator, Joaquim MATEO, MD, Hopital Lariboisière
Other Study IDs: JMATEO
Record Dates: First submitted 2018-11-16; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Radiography; Interventional

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: All monitoring — Dicpleth and PI are obtained a posteriori from the PPG waveform reconstruction and blindly from ABP values. Dicpleth is defined as the ratio of the height of the dicrotic notch (from nadir point of the complex to the notch) to the height of the systolic peak (from nadir point of the complex to the pic), measured at end-expiratory time (average of 3 consecutive complex). PI is calculated as the ratio of the pulsatile component of the PPG signal and the continuous component.

SUMMARY:
During general anaesthesia, intraoperative hypotension (IOH), defined as a mean arterial pressure (MAP) drop of more than 20%, is frequent with potential deleterious effects for patients. Pulse oximeter is mandatory in the operating room making photoplethysmographic (PPG) signal and parameters such as the relative dicrotic notch height (Dicpleth) or the perfusion index (PI) readily available. The purpose of this study is to investigate whether Dicpleth and PI could detect IOH during anaesthesia induction and follow their variations during vasopressor boluses.

DETAILED DESCRIPTION:
Main objective Haemodynamic stability is a major issue in the management of patients during general anaesthesia. Anaesthetic drugs induce rapid and deep systemic arterial blood pressure (ABP) drop which leads to intra operative hypotension (IOH) episodes. IOH can cause deleterious consequences such as myocardial infraction, cerebral hypoperfusion or acute kidney injury.

The major drawback of the oscillometric cuff is to measure ABP only at intermittent intervals. As ABP may vary quickly, especially during induction of anaesthesia, IOH should be detected in real time as even a short period of IOH may have deleterious consequences on vital organs.

Digital photoplethysmography (PPG) is a non-invasive signal produced by light absorption variations due to pulsatile blood volume variations. Indices derived from PPG signals have been used successfully to characterize cardiovascular state in patients.

Dicrotic notch height (Dicpleth), representing the relative height of the dicrotic wave compared to the maximum peak of the waveform, has been described as the amount of reflected wave, dependent of the vascular tone. Reduction in Dicpleth has been shown to be related to reduction of vascular tone due to vasodilator drugs such as salbutamol or glyceryl Trinitrate.

Perfusion Index (PI) represents the ratio of the pulsatile light absorption (i.e the amount of blood ejected at each systole) on the continuous absorption (corresponding to the non-pulsatile vessels, bones and soft tissues). PI has been described as a reliable tool for vascular tone assessment and monitoring

Primary Evaluation Criteria As Dicpleth and PI are both related to vascular tone and are easily derived from the PPG signal, Investigators aimed to explore whether the combined analysis of Dicpleth and PI variations would allow for early detection of IOH during the during a standardized propofol-remifentanil anesthesia induction.

Estimate the correlations between variations of Dicpleth and MAP, and PI and MAP during induction of anaesthesia and during bolus of vasopressors.

Estimate if a combined analysis of these two parameters enhanced diagnostic performance for detecting IOH under actions of vasoactive effect of anaesthetics.

Experimental design This is a single-center, interventional, category II prospective study (minimal risks and constraints) Population concerned The study involves major patients who beneficiate from intraoperative hemodynamic optimization with norepinephrine (as noradrenaline tartrate) for maintaining blood pressure under general anaesthesia in interventional neuroradiology in adults.

Research Proceedings Hemodynamic parameters (heart rate, systolic arterial pressure [SAP], mean arterial pressure [MAP] and diastolic arterial pressure [DAP]), and PPG parameters (Dicpleth, PI and SpO2) will be retrospectively sampled every minute during induction. All monitoring parameters and curves displayed on the monitor will be recorded on a computer with ixTrend© software (ixellence, Wildau, Germany). Investigators defined "pre-pressor" values as the measures prior to the vasopressor bolus during IOH episodes. "Peak-pressor" values is defined as the maximum effects of vasopressor bolus, when the highest MAP is reached. In agreement with most studies, IOH is defined as a MAP drop of more than 20% from baseline MAP.

In patients presenting a hypotensive episode, all parameters are collected before and at the peak effect of a 10µg bolus of norepinephrine

Individual benefit:

There is no benefit for the patient

Collective benefit:

As ABP may vary quickly, especially during induction of anaesthesia, IOH should be detected in real time as even a short period of IOH may have deleterious consequences on vital organs. The non-invasive combined analysis of Dicpleth and PI variations would allow for early detection of IOH during the induction of general anaesthesia.

Risks and minimal constraints added by the research No added risk This clinical research work is "non-interventional" on adult patients who benefit from a neuroradiological intervention. All measures are obtained non-invasively.

During their interventional neuroradiology procedure, all patients' routine monitoring will consist of electrocardiogram, pulsated oxygen saturation, end-tidal CO2, respiratory rate, tidal volume and monitoring of neuromuscular function.

For all patients whatever the comorbidities, anesthesia induction will be performed using a target-controlled infusion (Orchestra® Base Primea - Fresenius Kabi France).

In agreement with most studies, IOH is defined as a MAP drop of more than 20% from baseline MAP.

Hemodynamic parameters (heart rate, systolic arterial pressure [SAP], mean arterial pressure [MAP] and diastolic arterial pressure [DAP]), and PPG parameters (Dicpleth, PI and SpO2) will be retrospectively sampled every minute during induction.

In patients presenting a hypotensive episode, all parameters are collected before and at the peak effect of a 10µg bolus of norepinephrine.

Number of selected subjects The primary aim of the study is to estimate the AUC of the ROC curve of both ΔDicpleth and ΔPI to track IOH during induction. Sample size was determined with an expected AUC at 0.85, an expected incidence of hypotension of 80% and the width of the confidence interval of 1. With a power of 80%, the number of patients to include was then 62.15 Secondary objective is to evaluate AUC of the ROC curve for combination of ΔDicpleth and ΔPI.

Statistics Changes of the parameters are analysed using Wilcoxon rank test. Correlation tests between ΔDicpleth and ΔMAP in one hand, and ΔPI and ΔMAP are performed by using Spearman test. Areas under the curve (AUC) of Receiver Operating Characteristic (ROC) curve (with 95% confidence interval) of ΔDicpleth and ΔPI to detect IOH episode will be estimated and eventually compared using DeLong test. Youden method is used to determine the optimal ΔDicpleth and ΔPI cut-off values to detect IOH episodes. Values are expressed as median and interquartile range [25th;75th percentiles]. P<0.05 is considered as statistically significant. Statistical analysis is performed using Prism 6.00© (Graphpad Software, Inc, La Jolla, CA, USA) and R 3.3.0 software (R foundation for Statistical Computing, Vienna, Austria).

Patients who have non-measurable Dicpleth at baseline before induction of anaesthesia will be excluded from the analysis

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years, scheduled an elective interventional neuroradiology procedure requiring general anesthesia
* oral agreement obtained from each patient before anesthesia

Exclusion Criteria:

* age <18 years
* an emergency procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with scheduled an elective interventional neuroradiology procedure requiring general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-05-23 (Actual); Study Completion 2015-05-23 (Actual)

PRIMARY OUTCOMES:
Continuous measure of mean arterial pressure (MAP in mmHg) | Time Frame: duration of the interventional neuroradiology procedure: 1 day
  We calculated the variation of MAP during the induction period from the relative variations (in percent) from their baseline values. During vasopressor boluses, respective parameter's variations are calculated between "pre-pressor" and "peak-pressor" measurements.
Continuous measure of SpO2 in % by photoplethysmography | Time Frame: duration of the interventional neuroradiology procedure: 1 day
  We calculated variations of Dicpleth, and perfusion index (PI) during the induction period from the relative variations (in percent) from their baseline values. During vasopressor boluses, respective parameter's variations are calculated between "pre-pressor" and "peak-pressor" measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MATEO, MD, Principal Investigator — Hopital Lariboisière

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coutrot M, Joachim J, Depret F, Millasseau S, Nougue H, Mateo J, Mebazaa A, Gayat E, Vallee F. Noninvasive continuous detection of arterial hypotension during induction of anaesthesia using a photoplethysmographic signal: proof of concept. Br J Anaesth. 2019 May;122(5):605-612. doi: 10.1016/j.bja.2019.01.037. Epub 2019 Mar 11. PMID 30916032